CLINICAL TRIAL: NCT01527695
Title: A Phase IIA, Multi Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Effect of 8 Weeks Treatment With Oral AZD3241 on Microglia Activation, as Measured by Positron Emission Tomography (PET), in Patients With Parkinson's Disease
Brief Title: PET Study in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D0490C00004
Record Dates: First submitted 2011-12-22; First posted 2012-02-07 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
Keywords: Phase IIa; AZD3241; microglia activation; safety; Pharmacodynamics and pharmacokinetics analyses; Parkinson patients
MeSH Terms: conditions — Parkinson Disease | interventions — AZD3241

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD3241 (Experimental): AZD3241 tablets 25 mg or 100 mg, titration first 5 days (50 mg bd on Day 1, 100 mg bd on Day 2, 200 mg bd on Day 3, 300 mg bd on Day 4, 400 mg bd on Day 5) Maintenance treatment from Day 6, 600 mg bd until Day 56±3 days
  Interventions: Drug: ER tablet 25 mg AZD3241; Drug: ER tablet 100 mg AZD3241
- Placebo (Experimental): AZD3241 placebo bid for 8 weeks
  Interventions: Drug: Placebo for AZD3241 25 mg; Drug: Placebo for AZD3241 100 mg

INTERVENTIONS:
Drug: ER tablet 25 mg AZD3241 — 2 tablets twice daily for Day 1
  Arms: AZD3241
Drug: ER tablet 100 mg AZD3241 — 1-6 tablets twice daily from Day 2 until Day 56±3 days
  Arms: AZD3241
Drug: Placebo for AZD3241 25 mg — 2 tablets twice daily for Day 1
  Arms: Placebo
Drug: Placebo for AZD3241 100 mg — 1-6 tablets twice daily from Day 2 until Day 56±3 days
  Arms: Placebo

SUMMARY:
This is a multi-centre study to be conducted in Sweden and Finland. Up to 24 male and/or female patients of non-childbearing potential aged 45 to 75 years (inclusive), with a clinical diagnosis Parkinson's Disease will be randomised in the study to allow for 20 patients to complete this study.The study will evaluate the effect of 8 weeks treatment with AZD3241 on microglia activation as measured via PET examinations.

DETAILED DESCRIPTION:
A Phase IIA, Multi centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Effect of 8 Weeks Treatment with Oral AZD3241 on Microglia Activation, as Measured by Positron Emission Tomography (PET), in Patients with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged 45 to 75 years (inclusive) at the day of enrolment (Visit 1)
* Female patients must have a negative pregnancy test at Screening, must not be lactating and must be of non childbearing potential, confirmed at Screening
* Male patients should be willing to use barrier contraception, eg, condoms, even if their partners are post-menopausal, be surgically sterile or are using accepted contraceptive methods, from the administration of the first dose of the investigational
* The clinical diagnosis of patients must meet the criteria for "diagnosis of idiopathic Parkinson's disease" according to the modified UKPDS Brain Bank criteria (see Appendix E)
* Modified Hoehn and Yahr stage 1 to 2

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other Parkinsonian syndromes exists, such as secondary Parkinsonism (caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), Parkinson-plus syndromes or heredodegenerative diseases
* Patients who have undergone surgery for the treatment of Parkinson's disease (eg, pallidotomy, deep brain stimulation, foetal tissue transplantation) or have undergone any other brain surgery
* Presence of significant dyskinesias, motor fluctuations, swallowing difficulties or loss of postural reflexes Patients with a history of non-response (according to both the clinician and the patient) to an adequate course of L-dopa or a DA agonist
* Use of pergolide, selegiline, metoclopramide, strong CYP3A4 inhibitors, CYP3A4 inducers (including St John's Wort) and strong CYP1A2 inhibitors and inducers, within 1 month of randomisation;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change of binding [11C]PBR28 to translocator protein (TSPO) measured by Positron Emission Tomography (PET). | baseline, 2-4 weeks
Change of binding of [11C]PBR28 to TSPO measured by PET. | baseline, 7-8 weeks

SECONDARY OUTCOMES:
Adverse events, vital signs, electrocardiogram (ECG), physical examination, clinical chemistry tests, height and weight measures for safety and tolerability profile. | Up to 10 weeks
Change in plasma activity of myeloperoxidase (MPO). | baseline, up to 10 weeks
Plasma concentrations of AZD3241. | Up to 8 weeks
Part of safety profile in terms of Columbia Suicide Severity Rating Scale. | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Per Svenningsson, MD, PHD, Principal Investigator — Karolinska University Hospital; Bjorn Paulsson, MD, Study Director — AstraZeneca Medical Science Director
Locations (3):
- Sweden (3):
  - Reserach Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Vällingby